CLINICAL TRIAL: NCT01695187
Title: A Randomized, Double-Blind, Parallel-Group, Vehicle-Controlled, Multicenter Study of NB-001 Treatment of Recurrent Herpes Labialis
Brief Title: NB-001 Treatment of Recurrent Herpes Labialis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NanoBio Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NB-001-010
Record Dates: First submitted 2012-09-18; First posted 2012-09-27 (Estimated); Last update posted 2013-06-14 (Estimated); Status verified 2013-06

CONDITIONS: Herpes Labialis
Keywords: Herpes, Herpes Labialis, nanoemulsion, NanoBio, NB-001
MeSH Terms: conditions — Herpes Labialis; Herpes Simplex | interventions — 5-((2-(6-Amino-9H-purin-9-yl) ethyl) amino)-1-pentanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NB-001 (0.3%) (Experimental): NB-001 is an oil-in-water emulsion composed of nanometer-sized, positively charged droplets (average particle size = 180nm). NB-001 is composed of highly refined soybean oil, purified water, ethanol, edetate disodium dihydrate (EDTA) and two surfactants: polysorbate (Tween) 20 and cetylpyridinium chloride (CPC).
  Interventions: Drug: NB-001 (0.3%)
- Vehicle (Placebo Comparator): NB-001 is an oil-in-water emulsion composed of nanometer-sized, positively charged droplets (average particle size = 180nm). NB-001 is composed of highly refined soybean oil, purified water, ethanol, edetate disodium dihydrate (EDTA) and one surfactant: polysorbate (Tween) 20.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NB-001 (0.3%) — Topical administration at least five times throughout the day
  Arms: NB-001 (0.3%)
Drug: Placebo
  Arms: Vehicle

SUMMARY:
This is a study to test the hypothesis that time to healing of a cold sore will be lower in the active treatment arm of the study when compared to the vehicle (placebo). Subjects with a history of cold sores will be enrolled and administered active treatment or placebo in a blinded manner. Subjects will then be followed to assess time to healing.

ELIGIBILITY:
Inclusion Criteria:

1. Be a healthy man or woman 18 years of age or older. Women who are pregnant, lactating or may become pregnant may (at the investigator's discretion) be included in the study;
2. Have recurrent herpes labialis as defined by a history of three (3) or more cold sore recurrences on the lips and/or skin surrounding the lips in the previous year. The majority of their cold sore recurrences proceeded by a well-defined history of prodromal symptoms including redness, pain, burning, tingling, itching, swelling or a tight sensation of the lip at the site of the outbreak;
3. Be willing to refrain from using systemic or topical antiviral agents or systemic corticosteroids within 4 weeks prior to study drug administration and for the duration of the cold sore recurrence;
4. Be willing to refrain from using any topical pharmaceutical or cosmetic products other than the study medication in or around the nasal and perioral areas for the duration of the cold sore recurrence;
5. Be willing to refrain from participation in another clinical trial;
6. Be willing and able to use phone or internet to obtain the combination to unlock their study medication kit;
7. Be able to read and write in English and understand and comply with the protocol requirements;
8. Be able to give informed consent and have signed a written informed consent form.

Exclusion Criteria:

1. Known hypersensitivity to one of the drug ingredients, including soybean oil, polysorbate (Tween), alcohol, EDTA, or cetylpyridinium chloride (found in some mouthwashes and lozenges);
2. Severe chronic illness including renal failure, severe respiratory or cardiac disease, chronic infections, immunodeficiency syndrome, uncontrolled diabetes mellitus or untreated severe thyroid disease;
3. Received (within the last 6 months) or receiving chemotherapy;
4. Significant skin disease on the face (such as atopic dermatitis, cystic acne, severe rosacea, eczema, psoriasis or other chronic vesiculobullous disorders) or lesions, wounds, abrasions, piercings, tattoos, irritation or other skin conditions on or around the nasal and perioral areas that would interfere with the treatment or assessment of the primary lesion complex. Subjects with mild controlled psoriasis, eczema, acne or dermatitis or other conditions may be included if the condition does not interfere with the ability to evaluate a herpes labialis lesion or local skin irritation;
5. Previously received herpes vaccine;
6. Active alcohol or drug abuse;
7. Prior randomization into any NanoBio study;
8. Any condition that would potentially make them unable to participate for the entire trial period;
9. Known allergies to topical creams, ointments or other topical medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2012-10; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Time to healing of the primary lesion complex (in days or fraction thereof) as assessed by the investigator. | Time to healing will be assessed from treatment onset to resolution of symptoms (maximum of 16 days)
  Time to healing is the time from receiving the combination to unlock the medication and begin treatment to investigator assessed healing.

SECONDARY OUTCOMES:
Proportion of subjects in whom the primary lesion complex does not progress beyond the Papule/Edema Stage | Proportion of subjects in whom the primary lesion complex does not progress will be assessed from treatment onset to resolution of symptoms (maximum of 16 days)
  This analysis will be performed in the cohort of subjects whose primary lesion complex is assessed as being in the Prodrome (pain, burning, tingling, itching, redness, swelling, or a tight sensation of the lip), Erythema/Macule, Papule/Edema, or Aborted Stage by the investigator at the first post-treatment visit.

OTHER OUTCOMES:
Safety and tolerability | Safety and tolerability will be assessed from treatment onset to study close (expected average of 2 months)
  Safety and tolerability of NB-001 following topical administration as assessed by the number and severity of adverse events.

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Radiant Research, Inc, Chandler, Arizona
  - Radiant Research, Inc, Tucson, Arizona
  - Radiant Research, Inc. Chicago, Chicago, Illinois
  - Central Kentucky Research Associates, Inc., Lexington, Kentucky
  - Radiant Research, Inc., Edina, Minnesota
  - The Center for Pharmaceutical Research, P.C., Kansas City, Missouri
  - Radiant Research, Inc., St Louis, Missouri
  - Radiant Research, Inc., Anderson, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Research Across America, Dallas, Texas
  - Radiant Research, Inc., San Antonio, Texas
  - New River Valley Research Institute, Christiansburg, Virginia